CLINICAL TRIAL: NCT01270789
Title: A Randomized Controlled Study Assessing the Effect of Liraglutide on the Preservation of Beta-Cell Function in Patients With Type 2 Diabetes Mellitus: The LIraglutide and Beta-cell RepAir (LIBRA) Study
Brief Title: LIraglutide and Beta-cell RepAir (LIBRA) Study
Acronym: LIBRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0230-A
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes
Keywords: beta-cell function; GLP-1 analogue; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide administered as once daily sc injection
  Other Names: Victoza
  Arms: Liraglutide
Drug: placebo — placebo administered as once daily sc injection
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder characterized by progressive deterioration in the function of the pancreatic beta-cells, which are the cells that produce and secrete insulin (the hormone primarily responsible for the handling of glucose in the body). We propose a double-blind, randomized controlled study comparing the effect of liraglutide (a novel anti-diabetic drug with beta-cell protective potential) versus placebo, on the preservation of beta-cell function over one year in patients with T2DM. This study may demonstrate an important beta-cell protective capacity of liraglutide.

DETAILED DESCRIPTION:
In this study, patients with type 2 diabetes who meet randomization criteria will be randomized to either liraglutide or placebo, with serial assessment of beta-cell function over 48 weeks follow-up. The hypothesis under study is whether liraglutide can preserve beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

* men and women between the ages of 30 and 75 years inclusive
* physician-diagnosed type 2 diabetes of </= 7 years duration
* negative for anti-GAD antibodies
* on 0-2 oral anti-diabetic medications
* A1c at screening between 5.5% and 9.0% inclusive, if on oral anti-diabetic medications, or between 6.0% and 10.0% inclusive, if not on oral anti-diabetic medications

Exclusion Criteria:

* use of insulin, GLP-1 agonist, or dipeptidyl peptidase-4 (DPP-4) inhibitor
* type 1 diabetes or secondary forms of diabetes
* major illness with life expectancy < 5 years
* involvement in another study requiring drug therapy
* hypersensitivity to insulin, liraglutide, or metformin
* renal dysfunction
* hepatic dysfunction
* history of pancreatitis
* family or personal history of Multiple Endocrine Neoplasia type 2 (MEN-2) or familial medullary thyroid carcinoma
* personal history of non-familial medullary thyroid carcinoma
* malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
* excessive alcohol consumption
* unwillingness to undergo multiple daily insulin injection therapy
* unwillingness to perform capillary blood glucose monitoring at least 4 times per day during intensive insulin therapy
* congestive heart failure
* pregnancy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Preservation of beta-cell function measured by Insulin Secretion-Sensitivity Index-2 (ISSI-2) | 48-weeks
  ISSI-2 is a validated OGTT-derived measure of beta-cell function analogous to the disposition index obtained from the intravenous glucose tolerance test. ISSI-2 is defined as the product of (i) insulin secretion measured by the ratio of the area-under-the-insulin-curve (AUCins) to the area-under-the-glucose curve (AUCgluc) and (ii) insulin sensitivity measured by the Matsuda index.

SECONDARY OUTCOMES:
Glycemic Control | 48 weeks
  * A1c
  * Fasting glucose, 2 hour glucose, and AUCgluc on OGTT
  * Proportion of participants with A1c <7% at study end
  * Glucose tolerance status at study end (NGT, pre-diabetes, diabetes)
  * Proportion of participants with fasting glucose in non-diabetic range at study end (ie. <7.0 mmol/L)
  * Time to loss of glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Retnakaran, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nunez Lopez YO, Retnakaran R, Zinman B, Pratley RE, Seyhan AA. Predicting and understanding the response to short-term intensive insulin therapy in people with early type 2 diabetes. Mol Metab. 2019 Feb;20:63-78. doi: 10.1016/j.molmet.2018.11.003. Epub 2018 Nov 16. PMID 30503831
- [Derived] Kramer CK, Zinman B, Choi H, Connelly PW, Retnakaran R. Impact of the Glucagon Assay When Assessing the Effect of Chronic Liraglutide Therapy on Glucagon Secretion. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2729-2733. doi: 10.1210/jc.2017-00928. PMID 28472325
- [Derived] Kramer CK, Zinman B, Choi H, Retnakaran R. Predictors of sustained drug-free diabetes remission over 48 weeks following short-term intensive insulin therapy in early type 2 diabetes. BMJ Open Diabetes Res Care. 2016 Aug 1;4(1):e000270. doi: 10.1136/bmjdrc-2016-000270. eCollection 2016. PMID 27547422
- [Derived] Kramer CK, Zinman B, Choi H, Connelly PW, Retnakaran R. The Impact of Chronic Liraglutide Therapy on Glucagon Secretion in Type 2 Diabetes: Insight From the LIBRA Trial. J Clin Endocrinol Metab. 2015 Oct;100(10):3702-9. doi: 10.1210/jc.2015-2725. Epub 2015 Jul 31. PMID 26230296
- [Derived] Kramer CK, Zinman B, Choi H, Retnakaran R. Effect of Short-term Intensive Insulin Therapy on Post-challenge Hyperglucagonemia in Early Type 2 Diabetes. J Clin Endocrinol Metab. 2015 Aug;100(8):2987-95. doi: 10.1210/jc.2015-1947. Epub 2015 Jun 16. PMID 26079776
- [Derived] Stein CM, Kramer CK, Zinman B, Choi H, Opsteen C, Retnakaran R. Clinical predictors and time course of the improvement in beta-cell function with short-term intensive insulin therapy in patients with Type 2 diabetes. Diabet Med. 2015 May;32(5):645-52. doi: 10.1111/dme.12671. Epub 2015 Jan 7. PMID 25495067
- [Derived] Retnakaran R, Kramer CK, Choi H, Swaminathan B, Zinman B. Liraglutide and the preservation of pancreatic beta-cell function in early type 2 diabetes: the LIBRA trial. Diabetes Care. 2014 Dec;37(12):3270-8. doi: 10.2337/dc14-0893. Epub 2014 Sep 23. PMID 25249651
- [Derived] Kramer CK, Choi H, Zinman B, Retnakaran R. Glycemic variability in patients with early type 2 diabetes: the impact of improvement in beta-cell function. Diabetes Care. 2014 Apr;37(4):1116-23. doi: 10.2337/dc13-2591. Epub 2014 Feb 18. PMID 24550219
- [Derived] Kramer CK, Choi H, Zinman B, Retnakaran R. Determinants of reversibility of beta-cell dysfunction in response to short-term intensive insulin therapy in patients with early type 2 diabetes. Am J Physiol Endocrinol Metab. 2013 Dec 1;305(11):E1398-407. doi: 10.1152/ajpendo.00447.2013. Epub 2013 Oct 15. PMID 24129396